CLINICAL TRIAL: NCT03120325
Title: Therapeutic Potential and Neuroimmune Mechanisms of Vagal Nerve Stimulation on Gastrointestinal Motility and Inflammation
Brief Title: Vagal Nerve Stimulation for Gastroparesis
Acronym: VNS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges due to the COVID19 pandemic and funding not available to restart.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Linda Nguyen, Clinical Associate Professor, Medicine - Gastroenterology & Hepatology, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 39839
Record Dates: First submitted 2017-04-11; First posted 2017-04-19 (Actual); Results first posted 2023-04-05 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: 15 participants planned enrollment in each arm:
  * Diabetic Gastroparesis
  * Functional Dyspepsia
  * Idiopathic Gastoparesis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Idiopathic Gastroparesis (Experimental): Patients with idiopathic gastroparesis and delayed gastric emptying. All patients in trial will be giving themselves vagal nerve stimulation for two minutes on each side twice a day in the morning and the night for four weeks starting at visit 3 and ending at visit 5.
  Interventions: Device: Vagal Nerve Stimulation
- Diabetic Gastroparesis (Experimental): Patients with diabetic gastroparesis and delayed gastric emptying. All patients in trial will be giving themselves vagal nerve stimulation for two minutes on each side twice a day in the morning and the night for four weeks starting at visit 3 and ending at visit 5.
  Interventions: Device: Vagal Nerve Stimulation
- Functional Dyspepsia (Experimental): Patients with functional dyspepsia and normal gastric emptying. All patients in trial will be giving themselves vagal nerve stimulation for two minutes on each side twice a day in the morning and the night for four weeks starting at visit 3 and ending at visit 5.
  Interventions: Device: Vagal Nerve Stimulation

INTERVENTIONS:
Device: Vagal Nerve Stimulation — Patients will be giving themselves vagal nerve stimulation for four weeks at interval of two times a day for two minutes on each side for four weeks. The impact of the intervention on gastroparesis symptoms will be measured by upper endoscopy biopsies, blood work, autonomic function tests, survey data, stool samples, urine sample, and saliva samples before after after the four weeks of stimulation treatment.

SUMMARY:
This study is investigating a new form of treatment for a digestive disorder called gastroparesis. Gastroparesis is thought to be caused by a mix of inflammation and neural dysfunction. The vagal nerve is a large nerve originating from the brain that regulates digestive function. Patients with gastroparesis have what is a called a low vagal tone which results in gastrointestinal motility problems and inflammation; therefore, investigators hypothesize that increasing vagal tone through a hand-held vagal nerve simulator will reduce inflammation and gastrointestinal motility problems in gastroparesis patients. Investigators will evaluate this hypothesis through the use of upper endoscopy testing, breath testing, and blood, stool, urine, heart rate variability, and saliva testing before and after 4 weeks of vagal nerve stimulation (VNS) treatment.

There are 6 research visits

Visit 1 and visit 2 may take up to 8 weeks (screening/baseline) Visit 3 and visit 4 will take 4 weeks (VNS treatment) visit 5 and 6 will take approximately 4 weeks (VNS followup/washout)

Consequently, it is possible that if a patient were to be at the farthest ends of visit windows, they could potentially be in the study for approx 16 weeks. Visit 1 and 2 may be less than 8 weeks which would shorten the patient's overall involvement in the study.

The treatment phase of the study will always be 4 weeks with an additional 4 week washout phase.

Use of the VNS device takes 4 weeks. Endoscopy and blood work are taken before and after the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Age 21-65 years old.
3. Established diagnosis of functional dyspepsia, idiopathic or diabetic gastroparesis as per AGA (American Gastroenterology Association) guidelines.
4. Patient is capable of giving informed consent and undergo upper endoscopy.
5. Patient is on stable doses of other medications for gastroparesis for preceding 4 weeks prior to enrollment (baseline measures).

Exclusion Criteria

1. Surgical-related gastroparesis
2. Extrinsic myopathy or neuropathy causing gastroparesis.
3. Use of narcotic pain medications in the preceding 2 weeks of study enrollment.
4. Patients with enteric feeding tubes or requiring parenteral nutrition (Patients with g-tubes who are stable for 3 months and not using the g-tube for venting may be eligible. patient with J-tubes are not eligible.
5. Patients with severe flare requiring hospitalization.
6. Untreated significant depression or suicidal thoughts.
7. Pregnant or breast-feeding women.
8. History of gastric pacemaker implantation.
9. Patients with prior gastric surgery, including fundoplication, partial/total gastrectomy, or gastric bypass.
10. Patients with malabsorption of enteric, pancreatic, or hepatibiliary etiology.
11. Patients with primary pulmonary disorders that affect the spirulina breath test.
12. Patients with implantable electronic devices.
13. Patients with carotid artery atherosclerosis.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Gottfried, MD PHD, Principal Investigator — Stanford University; Linda Nguyen, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Idiopathic Gastroparesis: Patients with idiopathic gastroparesis and delayed gastric emptying self-administer vagal nerve stimulation for two minutes on each side twice a day in the morning and the night for four weeks (starting at visit 3 and ending at visit 5).
- Diabetic Gastroparesis: Patients with diabetic gastroparesis and delayed gastric emptying self-administer vagal nerve stimulation for two minutes on each side twice a day in the morning and the night for four weeks (starting at visit 3 and ending at visit 5).
- Functional Dyspepsia: Patients with functional dyspepsia and normal gastric emptying self-administer vagal nerve stimulation for two minutes on each side twice a day in the morning and the night for four weeks (starting at visit 3 and ending at visit 5).
Period: Overall Study
Arm/Group | Idiopathic Gastroparesis | Diabetic Gastroparesis | Functional Dyspepsia
Started | 17 | 1 | 6
Used Device (Received Treatment) | 15 | 1 | 5
Completed | 15 | 1 | 5
Not Completed | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Idiopathic Gastroparesis | Diabetic Gastroparesis | Functional Dyspepsia | Total
Number analyzed (Participants) | 15 | 1 | 5 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 1 | 5 | 21
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 1 | 4 | 18
  Male | 2 | 0 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 1 | 3 | 16
  Non-White | 3 | 0 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 1 | 5 | 21
Plasma cytokines [Mean (Standard Deviation); unit: Normalized mean fluoresc ent intensity] — Luminex assay median fluorescence intensity (MFI) data were preprocessed for each cytokine through a sequence of averaging over duplicate wells, natural-logarithm transformation to reduce variance heterogeneity, and isolation and the removal of plate effects. The average (mean) value across all cytokines is reported. Population: Data were not collected for the "Diabetic Gastroparesis" and "Functional Dyspepsia" groups.
  Normalized mean fluoresc ent intensity
    number analyzed (Participants) | 15 | 0 | 0 | 15
    (all) | 1 (0.3) |  |  | 1 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Vagal Nerve Stimulation on Gastroparesis Symptoms as Measures by the Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD) Questionnaire.
Description: Investigators will send daily GCSI-DD to patients for 8 weeks. This 10 item questionnaire measures the severity of gastroparesis symptoms on a scale 0-5. 0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, 5=very severe. Investigators hypothesize a change of more than 0.75 points. Scored were recorded daily at each time point and scores then averaged to produce an overall score (range: 0 to 5, higher scores correspond to worse symptoms).
Time Frame: Baseline (2 weeks prior to initiation), week 4 (7 days), week 8 (7 days)
Population: Participants who received treatment are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Idiopathic Gastroparesis | Diabetic Gastroparesis | Functional Dyspepsia
Number analyzed (Participants) | 15 | 1 | 5
score on a scale
  Baseline | 2.4 (0.76) | 2.68 (NA) — Standard deviation not calculable with an n of 1 | 2.1 (1.1)
  Week 4 | 1.65 (1.05) | 1.71 (NA) — Standard deviation not calculable with an n of 1 | 1.7 (1.0)
  Week 8 | 2.0 (1.09) | 2.36 (NA) — Standard deviation not calculable with an n of 1 | 1.6 (1.1)

2. Primary Outcome: Effect of Vagal Nerve Stimulation on the Gastric Emptying Spirulina Breath Test Emptying Time
Description: Investigators will measure a change in gastric emptying time before and after vagal nerve stimulation as measured in minutes. Higher number (longer times) indicate more severe gastroparesis.
Time Frame: Baseline and week 4 (3 hours to assess at each time point)
Population: Participants who received treatment are included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Idiopathic Gastroparesis | Diabetic Gastroparesis | Functional Dyspepsia
Number analyzed (Participants) | 15 | 1 | 5
minutes
  Baseline | 155.1 (40.2) | 140.8 (NA) — Standard deviation not calculable with an n of 1 | 91.8 (19.8)
  Week 4 | 129.0 (37.0) | 120.7 (NA) — Standard deviation not calculable with an n of 1 | 100.8 (37.7)

3. Secondary Outcome: PROMIS Pain Interference Questionnaire Score as a Measure of the Effect of VNS Therapy on Overall Pain
Description: The effect of VNS therapy on overall pain interference as assessed by the PROMIS (Patient Reported Outcomes Measurement Information System) pain interference questionnaire which is a 6 item questionnaire on a 5 point scale to assess the impact of pain on daily life. Scores are summed and converted to percentiles normalized for the population (normalized T-score). 50 indicates the population mean with a standard deviation of 10. The higher the T-score, the more severe the symptoms.
Time Frame: Baseline, week 4, week 8
Population: Participants who received treatment and with data at the respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Idiopathic Gastroparesis | Diabetic Gastroparesis | Functional Dyspepsia
Number analyzed (Participants) | 15 | 1 | 5
T-score
  Baseline | 64.5 (5.6) | 66.9 (NA) — Standard deviation not calculable with an n of 1 | 54.3 (8.0)
  Week 4 | 58.5 (7.9) | 65.5 (NA) — Standard deviation not calculable with an n of 1 | 58.8 (2.7)
  Week 8: number analyzed (Participants) | 15 | 0 | 5
  Week 8 | 63.6 (8.3) |  | 55.3 (10)

4. Secondary Outcome: Short Form 12 (SF-12) Score the Effect of VNS Therapy on Overall Wellbeing and Health
Description: The effect of VNS therapy on overall wellbeing and health as assessed by the SF-12. Score range: 0-100, higher scores correspond to better quality of life.
Time Frame: Baseline, week 4, week 8
Population: Participants who received treatment and with data at the respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Idiopathic Gastroparesis | Diabetic Gastroparesis | Functional Dyspepsia
Number analyzed (Participants) | 15 | 1 | 5
score on a scale
  Baseline | 64.2 (28.0) | 28.8 (NA) — Standard deviation not calculable with an n of 1 | 37.5 (8.4)
  Week 4 | 66.6 (29.7) | 37.7 (NA) — Standard deviation not calculable with an n of 1 | 44.1 (11.2)
  Week 8: number analyzed (Participants) | 15 | 0 | 5
  Week 8 | 63.1 (29) |  | 43 (10.8)

5. Secondary Outcome: Number of Participants With Any Serious or Treatment-emergent Adverse Event (AE) as a Measure of the Safety and Tolerability of VNS in Patients With Gastroparesis
Description: The safety and tolerability of VNS in patients with gastroparesis assessed by recording any side effects or adverse events. Number of patients reporting serious or treatment related adverse events are reported
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Idiopathic Gastroparesis | Diabetic Gastroparesis | Functional Dyspepsia
Number analyzed (Participants) | 17 | 1 | 6
Participants
  Serious AE | 0 | 0 | 0
  Treatment-emergent AE | 0 | 0 | 0

6. Secondary Outcome: Heart Rate Variability (HRV) as a Measure of the Effect of VNS Therapy on Vagal Tone
Description: The effect of VNS therapy on vagal tone as measured bv HRV (accounting for respiratory rate variability) using electrocardiogram (ASNAR) device. HRV is measured as an RFa value, a measure of the high-frequency heart rate (bpm^2 per hertz). Normal RFa is 0.5 to 8.0.
Time Frame: Baseline, week 4, week 8
Population: Participants who received treatment and with data at the respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: RFA (bpm^2/hertz)
Arm/Group | Idiopathic Gastroparesis | Diabetic Gastroparesis | Functional Dyspepsia
Number analyzed (Participants) | 15 | 1 | 5
RFA (bpm^2/hertz)
  Baseline | 10.6 (53.2) | 9.3 (NA) — Standard deviation not calculable with an n of 1 | 16.2 (36.7)
  Week 4 | 20.8 (84.0) | 2.2 (NA) — Standard deviation not calculable with an n of 1 | 11.2 (12.2)
  Week 8: number analyzed (Participants) | 15 | 0 | 5
  Week 8 | 25.1 (89.7) |  | 17.5 (25.5)

7. Secondary Outcome: Effect of VNS on Mucosal Inflammation
Description: Median fluorescence intensity (MFI) data were preprocessed for each cytokine through a sequence of averaging over duplicate wells, natural-logarithm transformation to reduce variance heterogeneity, and isolation and removal of plate effects. The effects of VNS therapy on gastric and small intestine inflammation was measured as average fold change across all tissue cytokines from endoscopic mucosal biopsies before and after VNS, using cytokine multiplex assays, which report relative levels of various cytokines as adjusted mean fluorescence intensity (MFI).
Time Frame: Baseline (pre-VNS) and 4 weeks (post-VNS)
Population: Participants who received treatment in the Idiopathic Gastroparesis group; data were not collected in the Diabetic Gastroparesis or Functional Dyspepsia groups.
Measure: Mean (Standard Deviation); unit: fold change of MFI
Units Other Than Participants: Cytokines
Arm/Group | Idiopathic Gastroparesis
Number analyzed (Participants) | 15
Number analyzed (Cytokines) | 53
fold change of MFI | 1 (0.01)

8. Secondary Outcome: The Effect of VNS Therapy on Gastric and Small Intestine Leukocyte Infiltration.
Description: The effects of VNS therapy on gastric and small intestine leukocyte infiltration was measured as relative abundance (normalized ratio) of immune cells (identified via CD45 marker) to total live cells across tissue leukocytes from endoscopic mucosal biopsies before and after VNS, using flow cytometry.
Time Frame: Baseline (pre-VNS) and 4 weeks (post-VNS)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: immune cell:total live cell ratio
Arm/Group | Idiopathic Gastroparesis
Number analyzed (Participants) | 15
immune cell:total live cell ratio
  Baseline | 0.76 (0.1)
  Week 4 | 0.76 (0.08)

ADVERSE EVENTS:
Time Frame: Baseline through week 8
Arm/Group | Idiopathic Gastroparesis | Diabetic Gastroparesis | Functional Dyspepsia
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/1 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/1 | 0/6
Other Adverse Events (participants affected / at risk) | 1/17 | 0/1 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idiopathic Gastroparesis (N=17) | Diabetic Gastroparesis (N=1) | Functional Dyspepsia (N=6)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
This trial had recruitment challenges due to the COVID19 pandemic with added cost of COVID testing prior to procedures. The idiopathic gastroparesis arm completed its planned enrollment but the other cohorts did not.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT03120325/Prot_SAP_000.pdf